CLINICAL TRIAL: NCT03929536
Title: Treatment of Acetabular Fractures in Elderly Patients
Acronym: ACETA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00520; ch19Saxer2
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Acetabular Fracture
Keywords: hip joint replacement; hip joint preserving surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study investigates surgical treatment of acetabular fractures in elderly patients (>60 years of age), either undergoing joint-preserving surgery or joint- replacement. 1 year- outcome with regard to mobility and autonomy is assessed.

ELIGIBILITY:
Inclusion Criteria:

* surgical treatment of acetabular fracture between 2009 and 2018

Exclusion Criteria:

* pathological fractures due to neoplasm or metastasis
* status after implantation of an endoprosthesis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acetabular fracture between 2009 and 2018 treated at the Department of Orthopedic and Trauma Surgery of University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Change in living arrangements | at baseline (right after surgery) and 1 year after surgery
  preservation of autonomy investigated by assessment of living arrangements: at home (by oneself, with a partner, with professional support), residential home for the elderly with occasional support, nursing home)

SECONDARY OUTCOMES:
number of rehospitalisations | single time point assessment 1 year after surgery
  number of rehospitalisations
number of re-surgeries | single time point assessment 1 year after surgery
  number of re-surgeries
mortality | single time point assessment 1 year after surgery
  number of deaths
infections | single time point assessment 1 year after surgery
  number and type of infections
Change in leg length difference | at baseline (right after surgery) and 1 year after surgery
  radiological leg length difference (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Saxer, Dr. med, Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland